CLINICAL TRIAL: NCT01104142
Title: Efficacy of Continuous Glucose Monitoring in Subjects With Type 1 Diabetes Mellitus on Multiple Daily Injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII) Therapy
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Andrew K. Balo/SVP, Clinical and Regulatory Affairs, and Quality Assurance, DexCom, Inc
Other Study IDs: PTL-900222
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MDI: Subject on multiple Daily Injections
  Interventions: Device: CGM
- CSII: Subjects on Continuous Subcutaneous Insulin Infusion
  Interventions: Device: CGM

INTERVENTIONS:
Device: CGM — Continuous Glucose Monitoring System

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Continuous Glucose Monitoring System (DexCom™ SEVEN PLUS®) and to evaluate the impact of CGM on glycemic control when worn for up to 6-months by subjects 18 to 70 years-old with Type 1 diabetes mellitus on MDI or CSII therapy.

The primary objective of this study is to demonstrate no statistically significant differences between MDI and CSII subjects in terms of A1C change at 6 months as compared to baseline. A secondary objective is to evaluate time spent outside of the euglycemic region (70 to 180 mg/dL) from the baseline (blinded month) to the conclusion of 6 month follow-up.

Safety data of the SEVEN PLUS System will also be collected and safety will be characterized by the incidence of Adverse Device Effects, Serious Adverse Device Events, and Unanticipated Adverse Device Effects experienced by study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years;
2. Have been diagnosed with Type 1 diabetes at least 3 years;
3. Have been treated on multiple daily injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII) insulin therapy for at last 6 months;
4. Willing not to switch method of insulin delivery (i.e., MDI to CSII, or CSII to MDI) while enrolled in this study;
5. Baseline A1C within 6.5% to 10.0% (may be determined by POC measurement, e.g., DCA 2000 to assess this inclusion criterion);
6. Patients on MDI should be on a stable dose of peak-less insulin (e.g., Lantus) once or twice a day along with any rapid acting prandial insulin analog (e.g., Humalog, Novolog, or Apidra);
7. Willing not to inject insulin or wear an insulin pump insertion set within 3 inches from the Sensor site during Sensor wear;
8. Willing to use only the blood glucose meter(s) provided to them for self-monitoring of blood glucose (SMBG) during Sensor wear;
9. Willing to take a minimum of 4 fingersticks per day during home use (2 for calibration purposes, 2 for comparative purposes);
10. Willing to refrain from the use of acetaminophen during the Sensor insertion period and for at least 24-hours prior to Sensor insertion;
11. Willing not to schedule a magnetic resonance (MRI) scan, computed tomography (CT) scan, or x-ray, for the duration of the study;
12. Able to speak, read, and write English.

Exclusion Criteria:

* 1. Have extensive skin changes/diseases that preclude wearing the Sensor on normal skin (e.g. extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites; 2. Subjects who have a known allergy to medical-grade adhesives; 3. Are pregnant as demonstrated by a positive pregnancy test within 72 hours of insertion or are planning to become pregnant during the course of study; 4. Have a hematocrit that is less than 30%, or greater than 55%; 5. Current participation in another investigational study protocol (if a subject has recently completed participation in another drug study, the subject must have completed that study at least 30 days prior to being enrolled in this study); 6. Have used CGM for 6 or more weeks (combined) during the 3 months prior to enrollment; 7. Have any condition that, in the opinion of the Investigator, would interfere with their participation in the trial or pose an excessive risk to study staff handling venous blood samples (e.g., known history of hepatitis B or C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical study population will consist of a minimum of 100, and up to 120 subjects with insulin-requiring diabetes mellitus on Multiple Daily Injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII) therapy; equal number of subjects will be enrolled among each therapy group. It is desirable to have a similar distribution of baseline A1C in each study group.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-04

CONTACTS AND LOCATIONS:
Overall Officials: Andrew K Balo, Study Chair — DexCom, Inc.
Locations (1):
- Barbara Davis Center for Childhood Diabetes, Aurora, Colorado, United States

REFERENCES:
- [Derived] Garg SK, Voelmle MK, Beatson CR, Miller HA, Crew LB, Freson BJ, Hazenfield RM. Use of continuous glucose monitoring in subjects with type 1 diabetes on multiple daily injections versus continuous subcutaneous insulin infusion therapy: a prospective 6-month study. Diabetes Care. 2011 Mar;34(3):574-9. doi: 10.2337/dc10-1852. Epub 2011 Jan 28. PMID 21278138